CLINICAL TRIAL: NCT03265912
Title: Evaluating a Novel Method of EEG Evoked Response Potential Analysis in Concussion Assessment - A GE Healthcare Companion Study: Advanced MRI Applications for Mild Traumatic Brain Injury-Phase 2 (mTBI-phase2)
Brief Title: Evaluating a Novel Method of EEG Evoked Response Potential Analysis in Concussion Assessment
Status: Completed | Type: Observational
Sponsor: ElMindA Ltd (Industry)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: ELM-36
Record Dates: First submitted 2017-08-20; First posted 2017-08-29 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Concussion, Mild; TBI (Traumatic Brain Injury); Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Mild Traumatic Brain Injury: Subjects enrolled in the GE healthcare study: Advanced MRI Applications for Mild Traumatic Brain Injury-Phase 2 (mTBI-phase 2), mTBI (Mild Traumatic Brain Injury) patient group also called as Arm 1 in this study.
- Non Mild Traumatic Brain Injury: Subjects enrolled in the GE healthcare study, Advanced MRI Applications for Mild Traumatic Brain Injury-Phase 2 (mTBI-phase 2), non-TBI (Non Mild Traumatic Brain Injury) patients also called as Arm 2 in this study.

SUMMARY:
mTBI is widely recognized as a major public health concern in the United States and worldwide. mTBI diagnosis remains a clinical challenge as no single test can diagnose every concussion. Recent advances in EEG evoked response potential analysis have led to a novel technique for assessing brain network activation (BNA) patterns. This study purpose is to study this BNA technology in individuals who have sustained a concussion.

DETAILED DESCRIPTION:
Mild traumatic brain injury (mTBI), also known as concussion, occurs commonly in sport and Motor Vehicle accidents. The Centers for Disease Control and Prevention estimate that as many as 3.8 million sport-related concussions occur annually in the United States. Despite ongoing research, there is no highly sensitive clinical test for cognitive function that can be rapidly applied in a sporting environment. This makes the clinical diagnosis of concussion particularly difficult, as the clinical presentation of concussion is highly variable with symptoms often evolving over time. Furthermore, with less than 10% of concussions resulting in loss of consciousness, self-reported symptom presence may be the only initial evidence of a concussion. These factors make concussion a challenging injury to diagnose. Given the variability in concussion presentations, there is no single test that can diagnose a concussion.

ElMindA, the sponsor of this study, has developed a novel method to automatically reveal functional networks of brain activity based on analysis of EEG Event Related Potential (ERP) data. This technological platform is capable of providing new metrics of brain function that can assist in patient evaluation and management. The analysis is done in two separate processes that are entirely separate and are performed independently of one another. Reference Brain Network Models of EEG data were recorded and analyzed from several groups of subjects to establish a set of group patterns that characterized the brain network activity of the group. EEG data from a single subject are processed to enable subject evaluation, as compared to the established group patterns. This individual analysis is the basis of the BNA scores computed for an individual subject.

Therefore, this investigation is designed to evaluate the clinical utility of ElMindA's BNA scores in detecting and managing concussive injuries.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in Arm 1 -mTBI group in the GE study: Advanced MRI Applications for Mild Traumatic Brain Injury-Phase 2 study
* Enrolled in Arm 2 -non TBI group in the GE study: Advanced MRI Applications for Mild Traumatic Brain Injury-Phase 2 study
* Males and females Aged 15-50
* Willingness to participate in the companion study and the ability to give informed assent (for children) and/or consent (for the parent of a minor or adults aged 18 years of age or older for themselves).

Exclusion Criteria:

* Hair types which might preclude appropriate scalp electrode cap fit. E.g: dread locks, corn rows etc.
* Significant sensory deficit e.g.: Deafness, and/or blindness
* Open scalp wound
* Active head lice infection

Ages: 15 Years to 50 Years | Sex: All
Age Groups: Child, Adult
Study Population: Adolescents, young adults and adults of both genders, enrolled in Advanced MRI Applications for Mild Traumatic Brain Injury-Phase 2 (mTBI-phase2) Age range: 15-50 years
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

PRIMARY OUTCOMES:
Assess the BNA database for Mild Traumatic Brain Injury and Non Mild Traumatic Brain Injury population. | This study duration is 12 months
  Functional networks of brain activity is measured using analysis of EEG Event Related Potential (ERP) data. Clinical assessments battery will be utilized in order to examine different sets of BNA database for Mild Traumatic Brain Injury and Non Mild Traumatic Brain Injury population.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Hospital for Special surery, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania